CLINICAL TRIAL: NCT02147158
Title: A Randomized, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Ulipristal Acetate for the Intermittent Treatment of Abnormal Uterine Bleeding Associated With Leiomyomas
Brief Title: A Study of the Efficacy and Safety of Ulipristal Acetate Intermittent Treatment for Abnormal Uterine Bleeding Associated With Leiomyomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UL1208
Record Dates: First submitted 2014-05-10; First posted 2014-05-26 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Leiomyoma; Uterine Hemorrhage
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- UPA 5 mg:Placebo (Experimental): Ulipristal Acetate (UPA) 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 2.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- UPA 10 mg:Placebo (Experimental): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 2.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- UPA 5 mg:UPA 5 mg (Experimental): UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily in both Treatment Course 1 and Treatment Course 2. There was a 2 menses drug-free interval in between courses.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- UPA 10 mg:UPA 10 mg (Experimental): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily in both Treatment Course 1 and Treatment Course 2. There was a 2 menses drug-free interval in between courses.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- Placebo:UPA 5 mg (Experimental): Matching placebo tablets (5 mg and 10 mg) orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 2.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo
- Placebo:UPA 10 mg (Experimental): Matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 2.
  Interventions: Drug: Ulipristal acetate (UPA); Drug: Placebo

INTERVENTIONS:
Drug: Ulipristal acetate (UPA) — Ulipristal acetate (UPA) tablet.
Drug: Placebo — Matching placebo tablet.

SUMMARY:
This study will evaluate the superiority of ulipristal acetate versus placebo for the treatment of abnormal uterine bleeding associated with uterine fibroids

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, 18-50 years, inclusive.
* Cyclic abnormal uterine bleeding (heavy or prolonged).
* Menstrual blood loss (MBL) of ≥ 80 mL as measured by the alkaline hematin method in the first 8 days of menses.
* Minimum of one discrete leiomyoma observable by transvaginal ultrasound.
* Endometrial biopsy without evidence of malignancy or atypical or non-atypical hyperplasia.

Exclusion Criteria:

* History of uterine surgery that would interfere with the study endpoints.
* Known coagulation disorder including bleeding disorder or clotting disorder.
* History of, or current uterine, cervix, ovarian, or breast cancer.
* Alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), or total bilirubin two times or greater than the upper limit of normal range.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females suffering with abnormal uterine bleeding associated with leiomyomas were treated in this study.
Enrollment: 432 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (63):
- United States (61):
  - Watson Investigational Site 138, Mesa, Arizona
  - Watson Investigational Site 147, Phoenix, Arizona
  - Watson Investigational Site 106, Scottsdale, Arizona
  - Watson Investigational Site 124, Tucson, Arizona
  - Watson Investigational Site 155, Little Rock, Arkansas
  - Watson Investigational Site 155, Encino, California
  - Watson Investigational Site 157, Hawaiian Gardens, California
  - Watson Investigational Site 134, La Mesa, California
  - Watson Investigational Site 127, San Diego, California
  - Watson Investigational Site 151, San Diego, California
  - Watson Investigational Site 159, Denver, Colorado
  - Watson Investigational Site 131, Clearwater, Florida
  - Watson Investigational Site 135, Miramar, Florida
  - Watson Investigational Site 132, North Miami, Florida
  - Watson Investigational Site 161, Orlando, Florida
  - Watson Investigational Site 123, Plantation, Florida
  - Watson Investigational Site 112, Sarasota, Florida
  - Watson Investigational Site 102, Wellington, Florida
  - Watson Investigational Site 101, West Palm Beach, Florida
  - Watson Investigational Site 160, Atlanta, Georgia
  - Watson Investigational Site 103, Sandy Springs, Georgia
  - Watson Investigational Site 117, Savannah, Georgia
  - Watson Investigational Site 113, Champaign, Illinois
  - Watson Investigational Site 119, Schaumburg, Illinois
  - Watson Investigational Site 162, Brownsburg, Indiana
  - Watson Investigational Site 104, Granger, Indiana
  - Watson Investigational Site 150, Covington, Louisiana
  - Watson Investigational Site 130, Metairie, Louisiana
  - Watson Investigational Site 116, New Orleans, Louisiana
  - Watson Investigational Site 108, Las Vegas, Nevada
  - Watson Investigational Site 107, Las Vegas, Nevada
  - Watson Investigational Site 111, Lawrenceville, New Jersey
  - Watson Investigational Site 158, Moorestown, New Jersey
  - Watson Investigational Site 115, Albuquerque, New Mexico
  - Watson Investigational Site 155, The Bronx, New York
  - Watson Investigational Site 126, Durham, North Carolina
  - Watson Investigational Site 128, Greensboro, North Carolina
  - Watson Investigational Site 145, New Bern, North Carolina
  - Watson Investigational Site 146, Raleigh, North Carolina
  - Watson Investigational Site 118, Winston-Salem, North Carolina
  - Watson Investigational Site 155, Cincinnati, Ohio
  - Watson Investigational Site 155, Cleveland, Ohio
  - Watson Investigational Site 148, Cleveland, Ohio
  - Watson Investigational Site 139, Englewood, Ohio
  - Watson Investigational Site 133, Philadelphia, Pennsylvania
  - Watson investigational site 142, Pittsburgh, Pennsylvania
  - Watson Investigational Site 105, West Reading, Pennsylvania
  - Watson Investigational Site 136, Bluffton, South Carolina
  - Watson Investigational Site 110, Charleston, South Carolina
  - Watson Investigational Site 153, Columbia, South Carolina
  - Watson Investigational Site 154, Greenville, South Carolina
  - Watson Investigational Site 155, Knoxville, Tennessee
  - Watson Investigational Site 122, Dallas, Texas
  - Watson Investigational Site 114, Frisco, Texas
  - Watson Investigational Site 109, Houston, Texas
  - Watson Investigational Site 155, Houston, Texas
  - Watson Investigational Site 120, San Antonio, Texas
  - Watson Investigational Site 129, Webster, Texas
  - Watson Investigational Site 152, Norfolk, Virginia
  - Watson Investigational Site 137, Virginia Beach, Virginia
  - Watson Investigational Site 121, Seattle, Washington
- Canada (2):
  - Watson Investigational Site 140, Hamilton, Ontario
  - Watson Investigational Site 144, Ottawa, Ontario

REFERENCES:
- [Derived] Coyne KS, Harrington A, Currie BM, Chen J, Gillard P, Spies JB. Psychometric validation of the 1-month recall Uterine Fibroid Symptom and Health-Related Quality of Life questionnaire (UFS-QOL). J Patient Rep Outcomes. 2019 Aug 23;3(1):57. doi: 10.1186/s41687-019-0146-x. PMID 31444600
- [Derived] Lukes AS, Soper D, Harrington A, Sniukiene V, Mo Y, Gillard P, Shulman L. Health-Related Quality of Life With Ulipristal Acetate for Treatment of Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):869-878. doi: 10.1097/AOG.0000000000003211. PMID 30969201
- [Derived] Liu JH, Soper D, Lukes A, Gee P, Kimble T, Kroll R, Mallick M, Chan A, Gillard P, Harrington A, Sniukiene V, Shulman LP. Ulipristal Acetate for Treatment of Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2018 Nov;132(5):1241-1251. doi: 10.1097/AOG.0000000000002942. PMID 30303900

RESULTS

PARTICIPANT FLOW:
Period: Treatment Course 1
Arm/Group | UPA 5 mg:Placebo | UPA 10 mg:Placebo | UPA 5 mg:UPA 5 mg | UPA 10 mg:UPA 10 mg | Placebo:UPA 5 mg | Placebo:UPA 10 mg
Started | 55 | 47 | 107 | 110 | 55 | 58
Completed | 51 | 38 | 99 | 97 | 49 | 50
Not Completed | 4 | 9 | 8 | 13 | 6 | 8
Not completed — Adverse Event | 1 | 4 | 3 | 4 | 1 | 2
Not completed — Lost to Follow-up | 2 | 4 | 3 | 3 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 1 | 1 | 5 | 3 | 2
Period: Off-Treatment Interval 1
Arm/Group | UPA 5 mg:Placebo | UPA 10 mg:Placebo | UPA 5 mg:UPA 5 mg | UPA 10 mg:UPA 10 mg | Placebo:UPA 5 mg | Placebo:UPA 10 mg
Started | 51 | 38 | 99 | 97 | 49 | 50
Completed | 41 | 34 | 84 | 82 | 41 | 45
Not Completed | 10 | 4 | 15 | 15 | 8 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 3 | 2 | 4 | 2
Not completed — Protocol Violation | 1 | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal of Consent | 4 | 3 | 5 | 10 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Other Miscellaneous Reasons | 2 | 0 | 3 | 2 | 0 | 0
Period: Treatment Course 2
Arm/Group | UPA 5 mg:Placebo | UPA 10 mg:Placebo | UPA 5 mg:UPA 5 mg | UPA 10 mg:UPA 10 mg | Placebo:UPA 5 mg | Placebo:UPA 10 mg
Started | 41 | 34 | 84 | 82 | 41 | 45
Completed | 40 | 29 | 79 | 77 | 41 | 43
Not Completed | 1 | 5 | 5 | 5 | 0 | 2
Not completed — Adverse Event | 0 | 4 | 2 | 1 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 1 | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0 | 1
Period: Off-Treatment Interval 2
Arm/Group | UPA 5 mg:Placebo | UPA 10 mg:Placebo | UPA 5 mg:UPA 5 mg | UPA 10 mg:UPA 10 mg | Placebo:UPA 5 mg | Placebo:UPA 10 mg
Started | 40 | 29 | 79 | 77 | 41 | 43
Completed | 36 | 25 | 69 | 66 | 39 | 39
Not Completed | 4 | 4 | 10 | 11 | 2 | 4
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 4 | 0 | 5 | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other Miscellaneous Reasons | 0 | 3 | 1 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | UPA 5 mg:Placebo | UPA 10 mg:Placebo | UPA 5 mg:UPA 5 mg | UPA 10 mg:UPA 10 mg | Placebo:UPA 5 mg | Placebo:UPA 10 mg | Total
Number analyzed (Participants) | 55 | 47 | 107 | 110 | 55 | 58 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (5.7) | 41.8 (5.2) | 40.9 (6.6) | 41.0 (5.3) | 40.8 (5.1) | 40.7 (4.6) | 41.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 47 | 107 | 110 | 55 | 58 | 432
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Bleeding During the Last 35 Consecutive Days on Treatment in Treatment Course 1
Description: Participants recorded bleeding in a daily diary. Absence of bleeding was defined as no bleeding days (i.e., no entries for bleeding or heavy bleeding; however, spotting was allowed), during the last 35 consecutive days on treatment in Treatment Course 1.
Time Frame: Last 35 consecutive days on treatment in the 12-Week Treatment Course 1
Population: Intent-to-Treat (ITT) Population included all randomized participants. Data was summarized as per the treatment assigned.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 1.
- UPA 5 mg: UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 1.
- UPA 10 mg: UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 1.
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 113 | 162 | 157
percentage of participants | 0.0 [0.0 to 3.8] | 42.0 [33.3 to 51.1] | 54.8 [45.5 to 63.8]

2. Primary Outcome: Time to Absence of Bleeding on Treatment During Treatment Course 1
Description: Time to absence of bleeding was defined as the duration in days from first dose to the first day in the time interval in which absence of bleeding occurs and persists through the last dose in the first treatment course. The persistence of absence of bleeding occurred for a minimum of 35 consecutive days counting backward from the last dose in Treatment Course 1.
Time Frame: From first dose up to the end of the 12-Week Treatment Course 1
Population: ITT population included all randomized participants. Data was summarized per treatment assigned.
Measure: Median (97.5% Confidence Interval); unit: days
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 113 | 162 | 157
days | NA [NA to NA] — Median and Confidence Interval (CI) were not estimable due to low number of participants with events. | NA [48.0 to NA] — Median and CI upper limit were not estimable due to low number of participants with events. | 36.0 [7.0 to NA] — CI upper limit was not estimable due to low number of participants with events.

3. Secondary Outcome: Percentage of Participants With Absence of Bleeding From Day 11 Through the End of Treatment Course 1
Description: Participants recorded bleeding in a daily diary. Absence of bleeding was defined as no bleeding days (i.e., no entries for bleeding or heavy bleeding; however, spotting was allowed), from Day 11 to the end of treatment in Treatment Course 1.
Time Frame: Day 11 through the end of treatment in the 12-Week Treatment Course 1
Population: ITT population included all randomized participants. Data was summarized as per the treatment assigned.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 113 | 162 | 157
percentage of participants | 0.0 [0.0 to 3.8] | 34.6 [26.3 to 43.5] | 55.4 [46.2 to 64.4]

4. Secondary Outcome: Percentage of Participants With Absence of Bleeding During the Last 35 Consecutive Days on Treatment in Treatment Course 2
Description: Participants recorded bleeding in a daily diary. Absence of bleeding was defined as no bleeding days (i.e., no entries for bleeding or heavy bleeding; however, spotting was allowed), during the last 35 consecutive days on treatment in Treatment Course 2.
Time Frame: Last 35 consecutive days on treatment in the 12-Week Treatment Course 2
Population: Data was summarized as per the treatment assigned. Number of participants analyzed are participants with data available for analysis at the given timepoint.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 2.
- UPA 5 mg: UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 2.
- UPA 10 mg: UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 2.
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 75 | 84 | 82
percentage of participants | 8.0 [2.6 to 17.9] | 40.5 [28.5 to 53.3] | 57.3 [44.4 to 69.6]

5. Secondary Outcome: Time to Absence of Bleeding on Treatment During Treatment Course 2
Description: Time to absence of bleeding is defined as the duration in days from first dose in treatment course 2 to the first day in the time interval in which absence of bleeding occurs and persists through the last dose in the second treatment course. The persistence of absence of bleeding occurred for a minimum of 35 consecutive days counting backward from the last dose in Treatment Course 2.
Time Frame: From first dose up to the end of treatment in the 12-Week Treatment Course 2
Population: Data was summarized as per treatment assigned. Number of participants analyzed are participants with data available for analysis at the given timepoint.
Measure: Median (97.5% Confidence Interval); unit: days
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 75 | 84 | 82
days | NA [NA to NA] — Median and CI were not estimable due to low number of participants with events. | NA [37.0 to NA] — Median and CI upper limit were not estimable due to low number of participants with events. | 7.5 [5.0 to NA] — CI upper limit was not estimable due to low number of participants with events.

6. Secondary Outcome: Change From Baseline in Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL) Revised Activities Subscale Score at the End of Treatment Course 1
Description: The UFS-QOL is a uterine fibroid-specific questionnaire consisting of 37 questions developed to evaluate symptoms of uterine fibroids and their impact on health-related quality of life in women with leiomyomas. The first 8 questions comprise the Symptom Severity subscale to assess symptoms experienced by women with uterine leiomyomas, the remaining 29 questions comprise 6 subscales (Concern, Activities, Energy/mood, Control, Self-consciousness, Sexual Function) which overall deal with women's feelings and experiences regarding impact of uterine leiomyoma symptoms on her life. Each item is scored between 1 and 5, where 1=none of the time or not at all and 5=all of the time or a very great deal. A Revised Activities subscale was created to include the most relevant items pertaining to physical and social activities with a total possible score of 0 to 100. Higher Revised Activities subscale scores indicate less impact on activities. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1-4) to End of 12-Week Treatment Course 1
Population: Data was summarized as per treatment assigned and included all participants with data at both Baseline and Week 12 in Treatment Course 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UPA 5 mg | UPA 10 mg
Number analyzed (Participants) | 95 | 146 | 132
score on a scale
  Baseline | 28.70 (24.56) | 27.52 (24.05) | 33.24 (27.00)
  Change from Baseline at Week 12 | 14.25 (28.77) | 50.19 (32.07) | 54.73 (32.32)

ADVERSE EVENTS:
Time Frame: From study drug administration in Treatment Course 1 until the end of the 12-week off-treatment follow-up period after Treatment Course 2 (Up to 42 weeks)
Description: Safety population included all participants who received study drug analyzed per treatment actually received. 1 patient randomized to UPA 5 mg:Placebo and 2 patients randomized to UPA 10 mg:Placebo actually received placebo in Treatment Course 1; are included in Placebo arm. 1 patient randomized to UPA 5 mg:Placebo actually received Placebo:UPA 5 mg; is included in Placebo:UPA 5 mg arm and 3 patients who received placebo in both courses are not included in safety analyses in Treatment Course 2.
Groups:
- Placebo (Treatment Course 1): Matching placebo tablets, orally, once daily for 12 weeks in Treatment Course 1. Includes AEs that occurred in Treatment Course 1 and the 2 menses drug-free interval.
- UPA 5 mg (Treatment Course 1): UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily in Treatment Course 1. Includes AEs that occurred in Treatment Course 1 and the 2 menses drug-free interval.
- UPA 10 mg (Treatment Course 1): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily in Treatment Course 1. Includes AEs that occurred in Treatment Course 1 and the 2 menses drug-free interval.
- UPA 5 mg:Placebo (Treatment Course 2): UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by placebo matching tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 2. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
- UPA 10 mg:Placebo (Treatment Course 2): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 2. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
- UPA 5 mg:UPA 5 mg (Treatment Course 2): UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily in both Treatment Course 1 and Treatment Course 2. There was a 2 menses drug-free interval in between courses. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
- UPA 10 mg:UPA 10 mg (Treatment Course 2): UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily in both Treatment Course 1 and Treatment Course 2. There was a 2 menses drug-free interval in between courses. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
- Placebo:UPA 5 mg (Treatment Course 2): Matching placebo tablets (5 mg and 10 mg) orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by UPA 5 mg tablet plus matching placebo 10 mg tablet, orally, once daily for 12 weeks in Treatment Course 2. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
- Placebo:UPA 10 mg (Treatment Course 2): Matching placebo tablets (5 mg and 10 mg), orally, once daily for 12 weeks in Treatment Course 1; followed by a 2 menses drug-free interval; followed by UPA 10 mg tablet plus matching placebo 5 mg tablet, orally, once daily for 12 weeks in Treatment Course 2. Includes AEs that occurred in Treatment Course 2 and 12 week follow-up.
Arm/Group | Placebo (Treatment Course 1) | UPA 5 mg (Treatment Course 1) | UPA 10 mg (Treatment Course 1) | UPA 5 mg:Placebo (Treatment Course 2) | UPA 10 mg:Placebo (Treatment Course 2) | UPA 5 mg:UPA 5 mg (Treatment Course 2) | UPA 10 mg:UPA 10 mg (Treatment Course 2) | Placebo:UPA 5 mg (Treatment Course 2) | Placebo:UPA 10 mg (Treatment Course 2)
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/161 | 0/155 | 0/40 | 0/33 | 0/84 | 0/82 | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/116 | 3/161 | 4/155 | 0/40 | 2/33 | 2/84 | 1/82 | 1/42 | 1/44
Other Adverse Events (participants affected / at risk) | 18/116 | 38/161 | 46/155 | 12/40 | 11/33 | 20/84 | 8/82 | 7/42 | 9/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Treatment Course 1) (N=116) | UPA 5 mg (Treatment Course 1) (N=161) | UPA 10 mg (Treatment Course 1) (N=155) | UPA 5 mg:Placebo (Treatment Course 2) (N=40) | UPA 10 mg:Placebo (Treatment Course 2) (N=33) | UPA 5 mg:UPA 5 mg (Treatment Course 2) (N=84) | UPA 10 mg:UPA 10 mg (Treatment Course 2) (N=82) | Placebo:UPA 5 mg (Treatment Course 2) (N=42) | Placebo:UPA 10 mg (Treatment Course 2) (N=44)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Treatment Course 1) (N=116) | UPA 5 mg (Treatment Course 1) (N=161) | UPA 10 mg (Treatment Course 1) (N=155) | UPA 5 mg:Placebo (Treatment Course 2) (N=40) | UPA 10 mg:Placebo (Treatment Course 2) (N=33) | UPA 5 mg:UPA 5 mg (Treatment Course 2) (N=84) | UPA 10 mg:UPA 10 mg (Treatment Course 2) (N=82) | Placebo:UPA 5 mg (Treatment Course 2) (N=42) | Placebo:UPA 10 mg (Treatment Course 2) (N=44)
Nausea (Gastrointestinal disorders) | 5 | 13 | 4 | 0 | 2 | 3 | 0 | 0 | 3
Fatigue (General disorders) | 5 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 8 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 7 | 16 | 0 | 2 | 5 | 1 | 3 | 1
Hot flush (Vascular disorders) | 2 | 12 | 18 | 0 | 0 | 5 | 4 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.